CLINICAL TRIAL: NCT00768742
Title: Clinical Study to Assess the Safety and Effectiveness of VizAblate(tm) Intrauterine Ultrasound-guided RF Ablation (IUUSgRFA) of Submucosal and Intramural Uterine Fibroids on the Reduction of Pictorial Blood Loss Assessment Scores
Brief Title: Safety and Effectiveness Study of RF Ablation of Uterine Fibroids to Reduce Menstrual Bleeding: the Fibroid Ablation Study
Acronym: FAST
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study revised and reinitiated under another protocol
Sponsor: Gynesonics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL00635; HC-126128
Record Dates: First submitted 2008-10-06; First posted 2008-10-08 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Leiomyoma; Uterine Fibroids; Menorrhagia
Keywords: Uterine Fibroid RF Ablation; Intrauterine Ultrasound; VizAblate
MeSH Terms: conditions — Leiomyoma; Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: VizAblate Intrauterine Ultrasound-Guided RF Ablation — VizAblate enables a minimally invasive procedure to visualize, target and treat uterine fibroids using ultrasound visualization and RF energy.

SUMMARY:
The primary objective of this study is to test the hypothesis that a minimum 75% volume radiofrequency ablation of fibroids associated with menorrhagia results in reduction of menstrual bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal
* Regular, consistent menstrual cycles
* Serum progesterone > 6 ng/ml (19 nmol/L)
* 2 months history of PBLAC score of 150-500
* Maximum of 4 type I, type II, or intramural fibroids
* Patient is at low risk for cervical cancer
* Hemoglobin > 6 g/dl
* Not at risk for pregnancy
* No desire for future fertility
* Willing and able to complete the follow-up requirements outlined in the study design section of the protocol
* Willing to sign a consent form

Exclusion Criteria:

* Subserosal fibroids.
* Any fibroid that obstructs access to the endometrial cavity
* FSH > 20 IU/L
* Pregnancy
* Evidence of disorders of hemostasis
* Use of GnRH agonist or depomedroxyprogesterone acetate or other implantable or injectable progestin and/or estrogen
* SERMS/SPRMS within the last 6 months
* Current use of any IUD or use of Mirena IUS within the last 3 months
* Gynecological malignancy or hyperplasia
* Known/suspected abdominal/pelvic cancer
* Active pelvic infection (e.g., active salpingitis or other pelvic inflammatory disease)
* Adenomyosis
* Previous surgical or ablative treatment for fibroids or menorrhagia
* Previous uterine artery embolization or occlusion
* Patient on anti-coagulation therapy
* Needing emergency surgery to treat fibroid symptoms
* Concomitant intrauterine polyps.
* Major medical or psychiatric illness affecting general health or patient's ability to comply with follow-up schedule or provide valid patient self-assessment data
* Contraindication to MRI
* Allergy to contrast media
* Mild renal insufficiency or worse
* Known renal disease
* Uncontrolled hypertension lasting 2 years or more
* Diabetes
* Uterine size > 10 weeks or 10 cm from ectocervix to fundus.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Menstrual bleeding as measured by the Pictorial Blood Loss Assessment Chart (PBLAC) | Baseline, 3 mo, 6 mo, 9 mo, 12 mo

SECONDARY OUTCOMES:
Rate of surgical reintervention | 12 mo
Quality of Life questionnaires | Baseline, 3 mo, 6 mo, 9 mo, 12 mo
Time required to return to normal daily activity | 7-14 days
Adverse events | At time of discharge, 7-14 days, 3 mo, 6 mo, 9 mo, 12 mo.
Subject tolerance of procedure rated via analog visual scale | Discharge
Fibroid dimension and non-perfused volume | Baseline, 1 day, 3 mo, 6 mo, 9 mo, and 12 mo
Pregnancy and pregnancy-related complications | 3 mo, 6 mo, 9 mo, and 12 mo

CONTACTS AND LOCATIONS:
Overall Officials: David Toub, M.D., Study Director — Gynesonics
Locations (3):
- Canada (3):
  - Victoria General Hospital; Mature Women's Centre, Winnipeg, Manitoba
  - Shirley E. Greenberg Women's Health Centre, The Ottawa Hospital, Ottawa, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario